CLINICAL TRIAL: NCT06870578
Title: Fostering Patient-oriented Research in Cardiometabolic Disease Pathogenesis and Prevention
Brief Title: Building Research for Intervention Development in Gliosis and Eating Habits
Acronym: BRIDGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ellen Schur, MD, MS, Professor: School of Medicine, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00020281; 2K24HL144917 (NIH)
Record Dates: First submitted 2025-02-28; First posted 2025-03-11 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Gliosis; Child Obesity; Eating
MeSH Terms: conditions — Gliosis; Pediatric Obesity | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Focus Group and Child Taste Test (Study 1) (No Intervention): No intervention is administered. Adult caregivers will participate in a focus group to assess feasibility of a controlled feeding study in children and children will complete a taste-test of a controlled feeding study menu.
- Study-provided food (Study 2) (Experimental): Participants will be provided all meals for a 7-day period. For the other 7-days of their enrollment, they will be asked to consume their usual diet.
  Interventions: Other: Diet modification
- Focus Group (Study 3) (No Intervention): No intervention is administered. Adult caregivers of children will participate in a focus group to learn from families about participating in research involving feeding studies in children.

INTERVENTIONS:
Other: Diet modification — In Study 2 only, children will be provided all meals for a 7-day period. Meals will consist of nutritious foods, calories provided will exceed the child's estimated daily caloric need, and children will be asked to consume meals ad libitum.
  Arms: Study-provided food (Study 2)

SUMMARY:
The goal of this study is to 1) use magnetic resonance imaging (MRI) to evaluate the effect of nutritious foods on inflammation in the human hypothalamus of children and 2) assess the feasibility and acceptability of nutritious food feeding intervention strategies in children with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

* Study1: Adult caregiver and Child age 9-11y. Willing to come to in-person focus group
* Study 2: Age 9-11y, BMI ≥85th and ≤95th percentile for age and sex
* Study 3:Adult caregiver with child who qualify for free or reduced-cost lunch in WA State. Child age 9-11y and with overweight.

Exclusion Criteria (study 1 child participants and study 3 criteria for children of adult participants):

* Significant health conditions including type 2 diabetes
* History of major weight loss or eating disorder
* Current use of medications known to alter appetite or body weight (e.g., stimulants for ADHD)
* Documented cognitive disorder
* Severe food allergies, vegetarian, or vegan (Study 1 only)
* Unable to make the session date

Exclusion Criteria (study 2, child participants):

* Significant health conditions including type 2 diabetes
* History of major weight loss or eating disorder
* Current use of medications known to alter appetite or body weight (e.g., stimulants for ADHD)
* Documented cognitive disorder
* MRI contraindication (e.g., braces, claustrophobia)
* Weight >330 pounds (MRI limit)
* Severe food allergies, vegetarian, or vegan
* Currently in formal weight loss program

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
T2 relaxation time by brain MRI | 7 days of diet intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Schur, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No